## **General Information**

| Primary Researcher(s): | Judith Tsui, Sara Glick, Emily Williams, Elizabeth Austin |
|---|---|
| Collaborators: | Alex Gojic, Andrea Radick |
| Project Title: | Evaluation of a community-pharmacy program for medications to treat and prevent HCV, opioid use disorders, overdose, and HIV among HCV-infected PWID. |
| Date: | July 11, 2022 |

# **Study Aims and Design**

### General Context / Purpose: A general context for the study and the particular contributions of the project

to autonomously perform testing and prescribing and dispensing medications.

The opioid epidemic is a major public health crisis in the United States, leading to substantial morbidity and mortality related to the consequences of opioid use disorders and injection drug use, namely hepatitis C virus (HCV), HIV, and overdose. Yet, we are at a unique historical moment, as we possess effective medications that can improve and sustain the lives of people who inject drugs (PWID). Currently there are medications that can be prescribed to 1) cure HCV (directly-acting antivirals or DAAs), 2) prevent HIV infection (Pre-exposure Prophylaxis [PrEP]), and 3) treat/prevent overdose (naloxone and medications to treat OUD). Furthermore, there is an unprecedented opportunity to eliminate HCV, a disease that is transmitted through injecting drugs. However, achieving the goals of elimination will require better systems for allowing PWID access to medications to cure hepatitis C, as well as medications to prevent overdose and HIV. Pharmacists and community-pharmacy programs may be an innovative solution for this problem. Collaborative Drug Therapy Agreements (CDTAs) allow pharmacists to have authority

## Aim(s): The objective(s) of the analysis

Aim 1: To conduct qualitative interviews with HCV-infected PWID to inform the development of a community-pharmacy program to expand access to medications to treat and prevent HCV, opioid use disorders, overdose, and HIV.

Aim 2: To pilot and evaluate a community-pharmacy program for medications to treat and prevent HCV, opioid use disorders, overdose, and HIV among HCV-infected PWID.

We will examine the following sub-aims:

1. The number/percent of participants who <u>successfully link to the community pharmacy program</u> and are seen for initial evaluation.

- 2. The number/percent who initiate medications for HCV.
- 3. Number/percent who receive other medications (naloxone, PrEP, and MOUD)
- 4. Baseline and 6-month follow-up substance use in past 30 days via modified Addiction Severity Index (ASI)
- 5. Baseline and 6-month follow-up the number of <u>injecting episodes using shared needle/syringe within the past 30 days</u> via the modified Risk Behaviors Survey (RBS)
- 6. Baseline and 6-month follow-up the number of episodes of unprotected vaginal or anal sex within the past 30 days via RBS
- 7. Self-reported participant Likert scale surveys of <u>satisfaction and willingness to refer an injecting partner to the community</u> pharmacy for treatment
- 8. The number/percent who complete treatment for HCV, defined as having received all planned medication doses.
- 9. SVR12 defined as undetectable HCV viral load at least 12-weeks post treatment completion

**NOTE:** This analysis plan does not include the data on injection network

Inclusion/Exclusion Criteria: Defines the population to be analyzed. Describe criteria that were part of original data collection and additional criteria needed for this particular project.

### **Inclusion criteria:**

- **1.** Age ≥18 years old
- 2. Injected any drug within the past 90 days (intravenous or intramuscular)
- 3. Tested positive for HCV (screening and/or confirmatory viral load) at a community testing site (syringe exchange programs, addiction treatment programs, homeless shelters, urban drop-in shelters and low-income housing sites)
- 4. HCV treatment naïve and not currently already receiving treatment
- 5. Willing to undergo evaluation for HCV at a community pharmacy

### **Exclusion criteria:**

- 1. People who plan to leave the Seattle area within 6 months
- 2. Do not wish to be treated for their HCV infection
- 3. Are known to be pregnant
- 4. Report impending incarceration that would disrupt clinical care
- 5. Are not comfortable reading and speaking English
- 6. Report being HIV-positive
- 7. Report having end-stage renal disease or require dialysis treatments
- 8. Report prior enrolled in (i.e. completed at least the initial intake appointment) the Kelley-Ross pharmacy program for hepatitis C treatment ("One Step Hep C Free")

# **Data and Variables Needed for Analysis**

Add rows to tables as needed

If a dataset or variable needs to be created / does not exist yet, you can note that here.

| Variable Name | Definition | Variable type | Sub-aim # |
|---|---|---|---|
| m6hcvtxpharmd | Since our first visit, were you seen by the pharmacist (refer to them by name) for hepatitis C medications? | Yes/no | 1 |
| ehrtxkelleyross,<br>ehrtxkrevaldoc (EHR) | Did this participant seek treatment through the KR community pharmacy program? (defined as presence of initial eval note by Kelley-Ross pharmacist) | Yes/no | 1 |

| Variable Name | Definition | Variable type | Sub-aim # |
|---|---|---|---|
| M6hcvpharmdmed | Since our first visit, did you take any medications to treat hepatitis C | yes/no | 2 |
| | through the <b>pharmacist</b> (Kathleen)? This can mean that you took only | | |
| | one pill, some of the pills, or all of the pills you were prescribed. | | |
| M6hcvpharmdmedcom pno | If no, why not? | Check all that apply | 2 |
| | Since our first visit, did you take any medications to treat hepatitis C | Yes/no | 2 |
| M6hcvothpromed | through the <b>provider</b> ? This can mean that you took only one pill, | | |
| | some of the pills, or all of the pills you were prescribed. | | |
| ehrtxinitiate (EHR) | Was treatment initiated? (Defined as meds were prescribed, | Yes/no | 2 |
| | regardless of showing up to receive) | | |
| | Why was treatment not initiated? | categorical | 2 |
| ehrtxwhynotinitiated | (Response options: ppt determined not appropriate for tx, ppt | | |
| (EHR) | verbalized not wanting tx, ppt never returned, ppt did not complete | | |
| | workup, other (check all that apply)) | | |
| M6hcvpharmdmedper<br>cent | On a scale of 0% to 100%, how much of your medication did you | Integer, 0-100 | 8 |
| | take? Where taking every pill would be 100%, taking half the pills | | |
| | would be 50% and not taking any pills would be 0%. If you are still in | | |
| | your hepatitis C treatment course, think about how much of the | | |
| | medications you should have taken to date. | | |

| M6hcvothpromedcom | Have you completed your treatment regimen for hepatitis C(normally | Yes/no | 8 |
|---|---|---|---|
| р | 8-12 weeks of daily medications)? | | |
| ehrtxinterrupt;<br>ehrothtxinterrupt<br>(EHR) | Does the EHR text mention a treatment interruption? | Yes/no | 8 |
| ehrtxinterruptdays,<br>ehrtxinterruptweek;<br>ehrothtxinterruptdays,<br>ehrothtxinterruptweek<br>(EHR) | If yes, how many days? And at what week did the interruption occur? | Integer, -100, 1-12 | 8 |
| ehrtxadherence (EHR) | Do the notes document non-adherence? | Yes/no | 8 |
| ehrtxdctx (EHR) | Did the provider pre-maturely discontinue treatment? | Yes/no | 8 |
| ehrrxreceived (EHR) | Did the participant ever pick-up/receive their medication from the pharmacist? | Yes/no | 8 |
| ehrrx1dispdate (EHR) | Date of first medication dispensation | Date_mdy | 8 |
| ehrrx2actualdispdate (EHR) | Date of actual second medication dispensation | Date_mdy | 8 |
| ehrrx3actualdispdate (EHR) | Date of actual third medication dispensation | Date_mdy | 8 |
| m6hcvpharmdsvr12 | Did you have a blood test to see if you were cured? | Yes/no | 9 |
| M6hcvothproccure | Has your provider told you that you are cured of hepatitis C? | Yes/no | 9 |
| m6hcvpharmdsvr12res<br>ult | What were the results of that test? | Categorical | 9 |
| ehrlabavailable (EHR) | Are there post treatment HCV viral load lab results? | Yes/no | 9 |
| ehrlabresultdetect,<br>ehrlabresultdetect2<br>(EHR) | Result (undetectable, detectable & quantifiable, detectable & unquantifiable) | Categorical | 9 |

# Descriptive/Other Variables of Interest (Baseline variables listed, 6-month follow-up variables start with "m6...":

| Variable Name | Definition | Variable type | Sub-aim # |
|---------------|------------|----------------------|-----------|
| age | Age | continuous | NA |
| race | race | Categorical, nominal | NA |

| hispanic | Ethnicity/Hispanic/latinx | Yes/no | NA |
|---|---|---|---|
| gendid | Gender identity | Categorical, nominal | NA |
| Shstay | In the past 90 days, or since [des_neg90daycalc_2], where have you typically spent the night? *read options to participant, check all that apply | Discrete, check all that apply | NA |
| Shemploy | How would you describe your current employment status? | Categorical, nominal | NA |
| shinsur | Do you currently have health insurance or health care coverage? | Yes/no | NA |
| shinsurtype | What kind of health insurance or coverage do you currently have? | Categorical, nominal | NA |
| txsought | Prior to participating in this study, have you ever sought treatment for hepatitis C? | Yes/no | NA |
| othrxhivpos | have ever been told that you are HIV-positive? | Yes/no | NA |
| othrxnalox | Do you currently have Naloxone (i.e. Narcan), a medication to treat<br>an overdose? It can be either on you right now, or at the place where<br>you stay. | Yes/no | 3 |
| othrxoudrx | In the past 12 months, since [des_neg1yearcalc], which of these medications have you been prescribed and used as directed? | Categorical, nominal | 3 |
| Othrxprepuse, or othrxprepnow | Have you ever used PrEP? Or taking now? | Yes/no | 3 |
| *asi | Variables for ASI substance use and injection drug use | ASI past 30 days<br>Route<br>Number of days | 4 |
| hivdayshare | How many times did you use a cooker/cotton/rinse water that had been used by another person who injects in the last 30 days? | Discrete, count<br>between 0-30 | 5 |
| hivshareafter | How many times did you share your works (needle/syringes) with somebody else after you used it in the last 30 days? | Discrete, count between 0-30 | 5 |
| Hivinsertvagcond<br>Hivinsertanalcond<br>Hivreceptvagcond<br>hivreceptanalcond | Episodes of sex without condom | Discrete, count<br>between 0-30 | 6 |
| M6pnexpplan | My navigator and I developed a plan for hepatitis C treatment. | Categorical, ordinal | 7 |
| M6pnexpunderstand | My navigator and I understand each other. | Categorical, ordinal | 7 |
| M6pnexpchange | We have established a good understanding of the kind of changes that would be good for me. | Categorical, ordinal | 7 |

| M6pnexpefficient | I believe the time my navigator and I are spending together is spent efficiently. | Categorical, ordinal | 7 |
|---|---|---|---|
| M6pnexpaccomp | My navigator understands what I am trying to accomplish. | Categorical, ordinal | 7 |
| M6pharmdexp | I had a positive experience with the pharmacist who saw me for hepatitis C. | Categorical, ordinal | 7 |
| M6pharmdexprecom | I would recommend the pharmacist to other people I know who inject drugs. | Categorical, ordinal | 7 |
| m6pharmdexpquest | The pharmacist addressed the healthcare concerns and questions that I brought up during our visit(s). | Categorical, ordinal | 7 |
| m6pharmdexphelp | The pharmacist was able to help me with the services I was seeking. | Categorical, ordinal | 7 |
| m6pharmdexpunderst and | The pharmacists were understanding of the difficulties I face trying to access healthcare. | Categorical, ordinal | 7 |
| m6pharmdexpwelcom<br>e | I felt welcomed in the setting where I saw the pharmacist. | Categorical, ordinal | 7 |

# **Analytic Plan**

### **Descriptive Analyses**

First we will calculate participant demographic and HCV treatment characteristics using their baseline survey data (see Table 1). Then Compare participant opioid use disorder (OUD) and PrEP medications, injection drug use practices, and HIV risk behavior characteristics at baseline and final visit (Table 2). Figure 1 shows a Diagram of participant progress from pre-enrollment to end of treatment. Figures 2 and 3 are stacked bar charts showing the participant responses on pharmacist care and patient navigator satisfaction Likert scale survey questions at the final visit.

## **Inferential Analyses**

McNemar's exact test for matched pairs or t-test to test for associations or difference in means between baseline and final visit (table 2).